CLINICAL TRIAL: NCT06405542
Title: EX-CIPN: An Exercise-based Rehabilitation Intervention to Treat Persistent Chemotherapy-Induced Peripheral Neuropathy (CIPN)
Brief Title: Exercise-based Rehabilitation to Treat Persistent Chemotherapy Induced Peripheral Neuropathy (CIPN)
Acronym: EX-CIPN
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-5839
Record Dates: First submitted 2024-05-02; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy
Keywords: Cancer Rehabilitation; Peripheral Neuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EX-CIPN Exercise- Based intervention (Experimental): This arm is provided with an intervention that includes an individualized exercise program, remote monitoring, and remote person-to-person clinical support.
  Interventions: Behavioral: EX-CIPN

INTERVENTIONS:
Behavioral: EX-CIPN — The 10-week intervention includes:
  Individualized Exercise Program: Each participant will receive an individualized progressive exercise program that includes cardiovascular and strength training as well as balance and desensitization exercises and will be adjusted to the needs of the patient.
  Remote Monitoring: Fitbit™ devices will be used to monitor patients' physical activity over the duration of the program. Fitness trackers can promote behaviour change and allows for self-monitoring and feedback to the participant.
  Remote Person-to-Person Clinical Support: Participants will have scheduled remote check-ins and health coaching sessions with their assigned RKin over Microsoft Teams (MSTeams) on weeks 2, 3, 4, 6, and 8 of the intervention. During these calls, the RKin will review, adapt, and progress the exercise program as needed, discuss and develop goals for the following week, and identify potential barriers and solutions in achieving their goals.

SUMMARY:
The goal of this clinical trial is to learn if the EX-CIPN exercise-based intervention is feasible, acceptable, and safe in participants with persistent chemotherapy-induced peripheral neuropathy (CIPN). It will also give insight on the effectiveness of the exercise intervention in treating CIPN symptoms. The main questions it aims to answer are:

* Is EX-CIPN safe, acceptable, and feasible in cancer survivors experiencing persistent CIPN?
* Are the study design and methods feasible (recruitment and retention rates, feasibility of data collection and procedures)?

Researchers will provide all participants with the exercise-based intervention.

Participants will:

* Complete assessments at baseline, immediately post-intervention, and 3-months post-intervention
* Complete a 10-week remote, individualized exercise program
* Receive health coaching calls on weeks 2, 3, 4, 6, and 8 of the intervention
* Wear a FitBit throughout the study to track physical activity and promote behaviour change

ELIGIBILITY:
Inclusion Criteria:

* Received a diagnosis of any cancer and treated with curative intent (no minimum dose) including Stage 3 & 4 gynecologic malignancies, treated in the platinum-sensitive setting
* Are > 6 months post-completion of chemotherapy (ie no other chemotherapeutic agents since completing of the chemotherapy regimen)
* Report > Grade 1 on the Patient Reported NCI Common Terminology Criteria for Adverse Events version 5.0 grading scale (numbness and tingling severity item) and neuropathic pain >3 on the Neuropathic Pain 4 (DN4) (interview) (0-7)
* The presence of peripheral neuropathy due to chemotherapy (following onset of chemotherapy), as established via clinical assessment
* May be on maintenance oncologic therapies (ie endocrine therapy, Poly (ADP-ribose) polymerase (PARP) inhibitors) not known to cause neuropathy
* No current plans for chemotherapy in the next 6 months
* Currently engaging in < 90min per week of planned moderate-intensity aerobic exercise
* Independent with ambulation and transfers with or without ambulatory assistance (EGOG 0-2)
* Able to communicate sufficiently in English to complete intervention, questionnaires, and consent
* Willing to participate in the intervention and attend in-person physical assessments
* Have access to and are able to operate videoconferencing.

Exclusion Criteria:

* Known neurological conditions influencing cognition and preventing safe or appropriate engagement with self-management and exercise recommendations
* Pre-existing neuropathy prior to the start of chemotherapy
* Are currently enrolled in other cancer rehabilitation or exercise-based programs/interventions.
* Are currently taking ado-trastuzumab emtansine (TDM1) (ex. Kadcyla)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-25 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Accrual Rate | Throughout study completion, up to 24 weeks.
  Assessed based on CONSORT criteria through a screening log that tracks data collected of all screened patients. Eligibility screening will be performed to identify eligible consented and eligible non-recruited individuals with non-recruitment reasons documented. Number of participants consented and enrolled will be tracked each month.
Retention Rates | Baseline, post-intervention (10 weeks), 3-months post-intervention (20-24 weeks)
  Retention rates will be calculated as the proportion of participants that attend each assessment time point. The investigators will also examine rates of complete and missing data.
Adherence | Through study completion, up to 24 weeks.
  Assessed through health coaching call attendance, Fitbit™ usage, and self-report completion of weekly exercise plan
Intervention Safety | Through study completion, up to 24 weeks.
  All adverse events will be scored on the CTCAE version 5.0 and documented during weekly appointments and at follow-up assessments with the Registered Kinesiologist (RKin). Assessment, tests, and all exercises will be stopped at any time if any pain or discomfort is experienced.

SECONDARY OUTCOMES:
Pain Intensity | Baseline, post-intervention (10 weeks), 3-months post-intervention (20-24 weeks)
  Measured using the numeric pain rating scale (NPRS). Scored on a 1-10 scale, 1 being no pain and 10 being worst pain imaginable.
CIPN Symptoms | Baseline, post-intervention (10 weeks), 3-months post-intervention (20-24 weeks)
  Measured using the European Organisation for Research and Treatment of Cancer Chemotherapy-Induced Peripheral Neuropathy (EORTC CIPN-20) questionnaire. Results are scored on a scale between 20-80 with higher scores meaning worse outcomes.
CIPN-related Disability | Baseline, post-intervention (10 weeks), 3-months post-intervention (20-24 weeks)
  Measured using the Rasch-built Overall Disability Scale for patients with chemotherapy-induced peripheral neuropathy CIPN-RODS. Results are scored on a scale between 0-56 with lower scores meaning worse outcomes.
Strength (Upper Body) | Baseline, post-intervention (10 weeks), 3-months post-intervention (20-24 weeks)
  Measured via handgrip dynamometry or grip strength test (GST).
Strength (Lower Body) | Baseline, post-intervention (10 weeks), 3-months post-intervention (20-24 weeks)
  Measured by a 30-second sit to stand test (30-s STS).
Balance | Baseline, post-intervention (10 weeks), 3-months post-intervention (20-24 weeks)
  Measured using the Short Physical Performance Battery (SPPB) Balance Test. The SPPB balance test provides a score from 0 to 4 with lower scores meaning worse outcomes.
Gait Speed | Baseline, post-intervention (10 weeks), 3-months post-intervention (20-24 weeks)
  Measured using the Four-Metre Gait Speed Test.
Aerobic Functional Capacity | Baseline, post-intervention (10 weeks), 3-months post-intervention (20-24 weeks)
  Measured using a 6-minute walk test (6MWT).

CONTACTS AND LOCATIONS:
Locations (1):
- ELLICSR: Health Wellness and Cancer Survivorship Centre, Toronto, Ontario, Canada